CLINICAL TRIAL: NCT05240586
Title: Pragmatic Randomized Controlled Trial of Pharmacopuncture Therapy for Cervical Disc Herniation: A Pilot Study
Brief Title: Pharmacopuncture Therapy for Cervical Disc Herniation: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Principal Investigator, In-Hyuk Ha, KMD, Director, Jaseng Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS-CT-2021-13
Record Dates: First submitted 2022-02-13; First posted 2022-02-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Cervical Disc Herniation
MeSH Terms: interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pharmacopunture therapy (Experimental): The physicians will choose the type and volume of pharmacopuncture according to participants' conditions.
  Interventions: Procedure: pharmacopuncture therapy
- acupuncture therapy (Active Comparator): The physicians will choose the type and number of acupuncture therapy according to participants' conditions.
  Interventions: Procedure: acupuncture therapy
- physical therapy, medication(prn) (Active Comparator): The physicians will choose the type and time of physical therapy according to participants' conditions. According to clinical judgment, clinicians can prescribe analgesics and muscle relaxants if necessary.
  Interventions: Procedure: physical therapy, medication(prn)

INTERVENTIONS:
Procedure: pharmacopuncture therapy — This is a pragmatic RCT, so the physicians will choose the type and volume of pharmacopuncture according to participants' conditions.
  Arms: pharmacopunture therapy
Procedure: acupuncture therapy — This is a pragmatic RCT, so the physicians will choose the type and number of acupuncture therapy according to participants' conditions.
  Arms: acupuncture therapy
Procedure: physical therapy, medication(prn) — This is a pragmatic RCT, so the physicians will choose the type and time of physical therapy according to participants' conditions. According to clinical judgment, clinicians can prescribe analgesics and muscle relaxants if necessary.
  Arms: physical therapy, medication(prn)

SUMMARY:
This is pilot study for a 3-arm parallel pragmatic randomized controlled trial that will compare pharmacopuncture therapy, acupunture therapy and physical therapy, medication(prn) for cervical disc herniation.

DETAILED DESCRIPTION:
This is a pragmatic RCT, so the physicians will choose the type and volume of pharmacopuncture, the type and number of acupuncture and the type and time of physical therapy according to participants' conditions, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of cervical disc herniation for less than 12 months
2. Numeric Rating Scale (NRS) of neck pain is more than 5
3. Symptoms of neuromuscular disease in one or both upper limbs (pain, pull, numbness, sensory abnormalities, motor abnormalities)
4. Discrimination findings above protusion, which can explain clinical symptoms on Cervical spine MRI or CT
5. 19-69 years old
6. participants who agreed and wrote informed consents

Exclusion Criteria:

1. Case of being diagnosed with a specific serious disease that may cause neck pain(Migration of cancer reaching to spine, acute fracture of spine, spine dislocation)
2. Progressive neurologic deficits or severe neurologic deficits
3. Cause of pain due to soft tissue disease, not the spine(Cancer, fibromyalgia, RA, goat, or etc.)
4. Other chronic diseases(stroke, MI, kidney disease, diabetic neuropathy, dimentia, epilepsy, or etc.) that may interfere with the interpretation of therapeutic effects or outcomes
5. Participants taking steroid, immunosuppressant, psychotropic medication, or taking other drugs that may affect outcomes
6. Inappropriate or unsafe pharmacopuncture therapy; hemorrhagic disease, taking anticoagulant drug, or severe diabetes patients who are likely to be infected
7. Participants who took NSAIDs or pharmacopuncture, acupuncture, physical therapy within 1 week
8. Pregnant, planning to get pregnant or lactating women
9. Participants who had undergone cervical surgery within 3 months
10. Participants who had participated in other clinical trial within 1 month, had participated in other study within 6 months from the date of selection, or have plan for participation in other trial during follow up period of this trial
11. Participants who can not write informed consent
12. Participants who is difficult to participate in the trial according to investigator's decision

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale (NRS) of neck pain | Week 1, 2, 3, 4, 5, 6, 7, 13, 25
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) of radiating arm pain | Week 1, 2, 3, 4, 5, 6, 7, 13, 25
  NRS is a pain scale in which the patient indicates their subjective pain as a whole number from 0 to 10, where 0 indicates 'no pain or discomfort' and 10 indicates 'the most severe pain and discomfort imaginable'.
Visual analogue scale (VAS) of neck pain and radiating arm pain | Week 1, 2, 3, 4, 5, 6, 7, 13, 25
  Visual analogue scale of radiating leg pain, minimum 0 to maximum 100, which is a higher score means a worse outcome.
Neck Disability Index (NDI) | Week 1, 7, 13, 25
  NDI is a functional disability questionnaire. The possible range of each item score is 0 to 5. Total score range is 0 (better outcome) to 100 (worse outcome).
Northwick Park Questionnaire (NPQ) | Week 1, 7, 13, 25
  NPQ measures the neck pain and the consequent patient disabilities. The questionnaire is divided in nine five-part sections. Each parameter is divided in five answer possibilities with points from 0 till 4. 0 is significant for no pain and 4 is significant for worst pain. The maximum score is 36 if all nine questions were answered and 32 if only the first eight questions were answered. The percentage ranges from 0% to 100%. The higher the percentage, the greater the disability and the pain.
Patient Global Impression of Change (PGIC) | Week 7, 13, 25
  Participants rate the improvement after treatment on a 7-point Likert scale (1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.)
Short Form-12 Health Survey version 2 (SF-12 v2) | Week 1, 7, 13, 25
  The SF-12 consists of 12 questions across 8 domains, and higher scores indicate better health-related quality of life.
EuroQol-5 Dimension (EQ-5D-5L) | Week 1, 7, 13, 25
  The EQ-5D-5L consists of 5 questions (mobility, self-care, usual activities, pain, anxiety/depression) that ask about the current state of health, and answers each question with 5 likert. (1=I have no problems about, 2=I have slight problems about, 3=I have moderate problems about, 4=I have severe problems about, 5=I am unable to about)

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, Ph.D., Study Director — Jaseng Medical Foundation
Locations (7):
- South Korea (7):
  - Kyung Hee University Korean Medicine Hospital, Seoul, Dongdaemun-gu
  - Kyung Hee University Korean Medicine Hospital at Gangdong, Seoul, Gangdong-gu
  - Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu
  - Bucheon Jaseng Hospital of Korean Medicine, Bucheon-si, Gyeonggi Province
  - Dongguk University Bundang Oriental Hospital, Seongnam-si, Gyeonggi-do
  - Haeundae Jaseng Hospital of Korean Medicine, Busan
  - Daejeon Jaseng Hospital of Korean Medicine, Daejeon